CLINICAL TRIAL: NCT05371158
Title: Patient-centered Development and Effectiveness of Online Acceptance and Commitment Therapy for Pain Interference in Cancer Survivors With Persistent Painful Chemotherapy-induced Neuropathy
Brief Title: Effectiveness of Online ACT for Pain Interference in Cancer Survivors With Chronic Painful CIPN
Acronym: QLIPP-CIPN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The trial was terminated early due to low participant enrollment. Over a period of 22 months, a total of 112 patients were recruited, with 57 randomly assigned to the ACT group and 55 to the WLC group.
Sponsor: Daniëlle van de Graaf (Other)
Collaborators: Dutch Cancer Society (Other); Comprehensive Cancer Centre The Netherlands (Other)
Responsible Party: Sponsor-Investigator, Daniëlle van de Graaf, PhD Candidate, Tilburg University
Organization: Tilburg University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12181
Record Dates: First submitted 2022-03-16; First posted 2022-05-12 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy; Cancer Survivors
Keywords: CIPN, cancer survivors, Acceptance and Commitment Therapy, eHealth, online, PROFILES registry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Online intervention (Experimental): The experimental condition includes an online psychological intervention with therapist email guidance based on Acceptance & Commitment Therapy (ACT). ACT is a form of Cognitive Behavioral Therapy, which focuses on acceptance of chronic pain in order to be able to perform valuable activities, instead of attempts of avoidance and controlling (Hayes et al., 2012). The main goal of ACT is increasing psychological flexibility, which includes the ability to act effectively according to personal values, with pain. ACT can thereby play a role in creating more realistic expectations regarding expectations of future pain relief. The intervention can be worked through in the participant's own living environment. It consists of 6 modules which can be worked through in 8 weeks.
  Interventions: Behavioral: Online intervention
- Control condition (No Intervention): The control condition includes a waiting list group that can receive treatment-as-usual. Participants are placed on a waiting list and receive the online psychological ACT intervention without email guidance directly after the first follow-up measurement. Participants placed on the waiting list will not receive the ACT intervention immediately. Participants do have the opportunity to access treatment as usual (TAU). Directly after the first, 3-month follow-up measurement these participants receive the opportunity to follow the intervention without email guidance by a therapist.

INTERVENTIONS:
Behavioral: Online intervention — The first module includes psychoeducation on neuropathic pain and CIPN (Table 1). Participants acquaintance themselves with intervention goals and mindfulness exercises central to ACT. In subsequent modules, participants learn about the aversive effects of pain avoidance, gain insight into their personal values, and work on pain acceptance. Participants exercise to recognize unhelpful thoughts about their pain and learn the difference between the subjective (judging) and objective self, and think about concrete actions to prevent relapse. The intervention primarily consists of text and experiential exercises, complemented with illustrations, metaphors and audio (mp3) files. Additional functionalities may be an outline of experiences by other CIPN patients and/or the ability to keep a diary. Participants in the experimental condition will receive therapist guidance.
  Other Names: Embrace Pain
  Arms: Online intervention

SUMMARY:
Rationale: An average of 30% of adult cancer survivors suffers from chemotherapy-induced peripheral neuropathy (CIPN) ≥ 6 months after completion of chemotherapy, and their quality of life (QoL) is strongly affected due to these symptoms. Treatment options are limited.

Objective: The goal of this study is to examine the effectiveness of an online psychological intervention based on Acceptance and Commitment Therapy (ACT) in a Randomized Controlled Trial (RCT) and compared to a treatment-as-usual control condition (TAU). We aim to improve pain interference in cancer survivors with chronic painful CIPN (present for at least 3 months) in the curative disease phase who were treated with chemotherapy treatment at least 6 months ago (irrespective of disease site).

Study design: It concerns a test of effectiveness of the ACT intervention in an RCT on quality of life. In total, 146 participants will be randomly allocated to one of two groups: the online ACT intervention with therapist email guidance or a control condition that receives treatment-as-usual. Patients in the control condition can follow the online ACT intervention directly after the 3 month-follow up measurement. Self-reported questionnaires will be conducted at baseline, after the intervention, and at 3- and 6-month follow-up. Additionally, interviews will be executed with a subgroup of interested patients afterwards, to explore intervention effects more in-depth. Participants will be sampled via various patient organizations, oncologists, and advertisements distributed via the PROFILES-registry that contains ongoing research projects on CIPN. Data will be collected online via the PROFILES-registry.

Study population: The population consists of adult cancer survivors in the curative disease phase suffering from painful CIPN for at least 3 months and who received chemotherapy treatment 6 or more months ago.

Intervention: An online ACT intervention was developed in the first phase of the QLIPP-CIPN study. In this study phase insights into daily limitations and quality of life of the patient population were gained, which served as the basis of the patient-centered development of the online ACT intervention following the CeHRes roadmap for participatory eHealth design. The intervention includes an 8-week self-management course containing 6 modules regarding psycho-education and ACT- processes. By means of text and exercises people learn to carry out value-oriented goals in daily life with pain. To do this, they learn new ways of coping with pain, including reducing pain avoidance and increasing pain acceptance. Additionally, participants will receive email guidance.

Main study parameters/endpoint: Pain interference in daily life using subscale Interference of the Multidimensional Pain Inventory (MPI). This scale focuses on a psychosocial aspect of chronic pain, specifically the interference with functioning in, for example, work, homework chores, recreational and social activities due to pain.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Participation is not expected to have any risks. Participants can quit the study at any moment and will not be excluded based on medication use or other current treatment for CIPN. If participants regress during the intervention and need new chemotherapy treatment, they can choose if they will continue or not. Participants do need to invest time to follow the intervention, which takes around 2 hours per week. Furthermore, it might be confronting to work on pain acceptance for participants. Benefits of participation are foremost a possible improvement in pain interference and reductions in pain and CIPN symptoms.

ELIGIBILITY:
Inclusion criteria:

1. age of 18 years or older,
2. identified by a clinician or self as having painful sensations (i.e., aching, burning, ''pins-and-needles'', shock-like, painful tingling, numbness, cramps) bilaterally in the feet/legs and/or hands/arms for at least 3 months. Furthermore,
3. score a 3 or higher on an 11-point pain intensity scale (Numeric Rating Scale),
4. the pain was not present prior to receiving chemotherapy,
5. chemotherapy ended at least 6 months ago.

Exclusion criteria:

1. enrollment in psychological treatment related to cancer, pain, or psychiatry upon entry,
2. new chemotherapy scheduled during study participation,
3. no access to the Internet/no email address,
4. not enough time to follow the intervention (2 hours per week),
5. problems with the Dutch language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Pain interference | T0b (0 months)
  Multidimensional Pain Inventory - Dutch Language Version (MPI-DLV). Subscale Interference. Minimum = 0, maximum = 60. Higher score means worse outcome.
Pain interference | T1 (3 weeks)
  Multidimensional Pain Inventory - Dutch Language Version (MPI-DLV). Subscale Interference. Minimum = 0, maximum = 60. Higher score means worse outcome.
Pain interference | T2 (6 weeks)
  Multidimensional Pain Inventory - Dutch Language Version (MPI-DLV). Subscale Interference. Minimum = 0, maximum = 60. Higher score means worse outcome.
Pain interference | T3 (2 months)
  Multidimensional Pain Inventory - Dutch Language Version (MPI-DLV). Subscale Interference. Minimum = 0, maximum = 60. Higher score means worse outcome.
Pain interference | T4 (5 months)
  Multidimensional Pain Inventory - Dutch Language Version (MPI-DLV). Subscale Interference. Minimum = 0, maximum = 60. Higher score means worse outcome.
Pain interference | T5 (8 months)
  Multidimensional Pain Inventory - Dutch Language Version (MPI-DLV). Subscale Interference. Minimum = 0, maximum = 60. Higher score means worse outcome.

SECONDARY OUTCOMES:
Cancer related quality of life | T0b (0 months)
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaires Core-30 item (EORTC QLQ-C30). Minimum = 30, maximum = 126. Higher score means better outcome.
Cancer related quality of life | T3 (2 months)
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaires Core-30 item (EORTC QLQ-C30). Minimum = 30, maximum = 126. Higher score means better outcome.
Cancer related quality of life | T4 (5 months)
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaires Core-30 item (EORTC QLQ-C30). Minimum = 30, maximum = 126. Higher score means better outcome.
Cancer related quality of life | T5 (8 months)
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaires Core-30 item (EORTC QLQ-C30). Minimum = 30, maximum = 126. Higher score means better outcome.
CIPN symptom severity | T0a (0 months)
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-CIPN20 (EORTC QLQ-CIPN20). Minimum = 0, maximum = 60. Higher score means worse outcome.
CIPN symptom severity | T3 (2 months),
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-CIPN20 (EORTC QLQ-CIPN20). Minimum = 0, maximum = 60. Higher score means worse outcome.
CIPN symptom severity | T4 (5 months)
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-CIPN20 (EORTC QLQ-CIPN20). Minimum = 0, maximum = 60. Higher score means worse outcome.
CIPN symptom severity | T5 (8 months)
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-CIPN20 (EORTC QLQ-CIPN20). Minimum = 0, maximum = 60. Higher score means worse outcome.
Pain intensity | T0a (0 months)
  Numeric Rating Scale (NRS-11). Minimum = 0, maximum = 20. Higher score means worse outcome.
Pain intensity | T3 (2 months)
  Numeric Rating Scale (NRS-11). Minimum = 0, maximum = 20. Higher score means worse outcome.
Pain intensity | T4 (5 months)
  Numeric Rating Scale (NRS-11). Minimum = 0, maximum = 20. Higher score means worse outcome.
Pain intensity | T5 (8 months)
  Numeric Rating Scale (NRS-11). Minimum = 0, maximum = 20. Higher score means worse outcome.
Pain catastrophizing | T0b (0 months)
  Pain Catastrophizing Scale (PCS). Minimum = 0, maximum = 65. Higher score means worse outcome.
Pain catastrophizing | T1 (3 weeks)
  Pain Catastrophizing Scale (PCS). Minimum = 0, maximum = 65. Higher score means worse outcome.
Pain catastrophizing | T2 (6 weeks)
  Pain Catastrophizing Scale (PCS). Minimum = 0, maximum = 65. Higher score means worse outcome.
Pain catastrophizing | T3 (2 months)
  Pain Catastrophizing Scale (PCS). Minimum = 0, maximum = 65. Higher score means worse outcome.
Pain catastrophizing | T4 (5 months)
  Pain Catastrophizing Scale (PCS). Minimum = 0, maximum = 65. Higher score means worse outcome.
Pain catastrophizing | T5 (8 months)
  Pain Catastrophizing Scale (PCS). Minimum = 0, maximum = 65. Higher score means worse outcome.
Psychological distress | T0b (0 months)
  Hospital Anxiety and Depression Scale (HADS). Minimum = 0, maximum = 56. Higher score means worse outcome.
Psychological distress | T1 (3 weeks)
  Hospital Anxiety and Depression Scale (HADS). Minimum = 0, maximum = 56. Higher score means worse outcome.
Psychological distress | T2 (6 weeks)
  Hospital Anxiety and Depression Scale (HADS). Minimum = 0, maximum = 56. Higher score means worse outcome.
Psychological distress | T3 (2 months)
  Hospital Anxiety and Depression Scale (HADS). Minimum = 0, maximum = 56. Higher score means worse outcome.
Psychological distress | T4 (5 months)
  Hospital Anxiety and Depression Scale (HADS). Minimum = 0, maximum = 56. Higher score means worse outcome.
Psychological distress | T5 (8 months)
  Hospital Anxiety and Depression Scale (HADS). Minimum = 0, maximum = 56. Higher score means worse outcome.
Psychological flexibility | T0a (0 months)
  Psychological Inflexibility in Pain Scale (PIPS). Minimum = 0, maximum = 84. Higher score means worse outcome (higher score means more inflexibility).
Psychological flexibility | T1 (3 weeks)
  Psychological Inflexibility in Pain Scale (PIPS). Minimum = 0, maximum = 84. Higher score means worse outcome (higher score means more inflexibility).
Psychological flexibility | T2 (6 weeks)
  Psychological Inflexibility in Pain Scale (PIPS). Minimum = 0, maximum = 84. Higher score means worse outcome (higher score means more inflexibility).
Psychological flexibility | T3 (2 months)
  Psychological Inflexibility in Pain Scale (PIPS). Minimum = 0, maximum = 84. Higher score means worse outcome (higher score means more inflexibility).
Psychological flexibility | T4 (5 months)
  Psychological Inflexibility in Pain Scale (PIPS). Minimum = 0, maximum = 84. Higher score means worse outcome (higher score means more inflexibility).
Mindfulness | T0b (0 months)
  Freiburg Mindfulness Inventory (FMI). Minimum = 0, maximum = 56. Higher score means better outcome.
Mindfulness | T1 (3 weeks)
  Freiburg Mindfulness Inventory (FMI). Minimum = 0, maximum = 56. Higher score means better outcome.
Mindfulness | T2 (6 weeks)
  Freiburg Mindfulness Inventory (FMI). Minimum = 0, maximum = 56. Higher score means better outcome.
Mindfulness | T3 (2 months)
  Freiburg Mindfulness Inventory (FMI). Minimum = 0, maximum = 56. Higher score means better outcome.
Mindfulness | T4 (5 months)
  Freiburg Mindfulness Inventory (FMI). Minimum = 0, maximum = 56. Higher score means better outcome.
Mindfulness | T5 (8 months)
  Freiburg Mindfulness Inventory (FMI). Minimum = 0, maximum = 56. Higher score means better outcome.
Values-based living | T0b (0 months)
  Engaged Living Scale (ELS). Minimum = 0, maximum = 80. Higher score means better outcome.
Values-based living | T1 (3 weeks)
  Engaged Living Scale (ELS). Minimum = 0, maximum = 80. Higher score means better outcome.
Values-based living | T2 (6 weeks)
  Engaged Living Scale (ELS). Minimum = 0, maximum = 80. Higher score means better outcome.
Values-based living | T3 (2 months)
  Engaged Living Scale (ELS). Minimum = 0, maximum = 80. Higher score means better outcome.
Values-based living | T4 (5 months)
  Engaged Living Scale (ELS). Minimum = 0, maximum = 80. Higher score means better outcome.
Values-based living | T5 (8 months)
  Engaged Living Scale (ELS). Minimum = 0, maximum = 80. Higher score means better outcome.
Intervention evaluation (Based on: Trompetter et al. (2015)). | T3 (2 months) (ACT)
  Questions:
  * During the past few weeks, how many hours did you spend on average per week working on the online course?
  * On average, how many days per week did you do mindfulness exercises during the past few weeks?
  * On the days you practiced mindfulness: On average, how many minutes did you spend practicing?
  * How do you rate the quality of the online training you received?
  * Did you receive the kind of help you were hoping to receive?
  * To what extent did the online training meet your needs?
  * Suppose one of your acquaintances needed the same help, would you recommend the online training?
  * How satisfied are you with the amount of help you received?
  * Did the online training help you cope better with your problems?
  * Overall, how satisfied are you with the online training you received?
  * Would you do the online training again if you needed to?
  * What grade would you give the online training?
Intervention evaluation (Based on: Trompetter et al. (2015)). | T5 (8 months) (WLC)
  Questions:
  * During the past few weeks, how many hours did you spend on average per week working on the online course?
  * On average, how many days per week did you do mindfulness exercises during the past few weeks?
  * On the days you practiced mindfulness: On average, how many minutes did you spend practicing?
  * How do you rate the quality of the online training you received?
  * Did you receive the kind of help you were hoping to receive?
  * To what extent did the online training meet your needs?
  * Suppose one of your acquaintances needed the same help, would you recommend the online training?
  * How satisfied are you with the amount of help you received?
  * Did the online training help you cope better with your problems?
  * Overall, how satisfied are you with the online training you received?
  * Would you do the online training again if you needed to?
  * What grade would you give the online training?
Adherence | T5
  Adherence will be based on technical data obtained from Karify's online environment. The following information will be used for this purpose.
  * Sent messages: the moment when a message is sent to the supervisor.
  * Given feedback: the moment when feedback is given on a specific assignment.
  * Significant moment: first_viewed: the moment when an assignment is viewed for the first time.
  * Significant moment: finished: the moment when an assignment is handed in for the first time.
  This will possibly be combined with the number of hours spent on intervention (self-reported), as described under 'intervention evaluation'.

OTHER OUTCOMES:
Interviews | T3 (2 months)
  Qualitative data on intervention effects and satisfaction will be collected by means of interviews with some participants after completion of the intervention
Interviews | T5 (8 months)
  Qualitative data on intervention effects and satisfaction will be collected by means of interviews with some participants after completion of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Floortje Mols, PhD, Principal Investigator — Tilburg University
Locations (1):
- Tilburg University, Tilburg, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
PROFILES data is freely available (FAIR principles) for non-commercial scientific research trough www.profilesregistry.nl.
Supporting Information: Study Protocol
Time Frame: Data will be stored in a secure location (PROFILES registry) for 15 years.
Access Criteria: Raw data from the PROFILES registry is available for non-commercial scientific research, subject to study question, privacy, and confidentiality restrictions, and registration.
URL: http://www.profilesregistry.nl

REFERENCES:
- [Background] Hayes, S. C., Strosahl, K., and Wilson, K. G. (2012) Acceptance & Commitment Therapy: The process and practice of mindful change 2nd. Guilford Press.
- [Background] van de Poll-Franse LV, Horevoorts N, Schoormans D, Beijer S, Ezendam NPM, Husson O, Oerlemans S, Schagen SB, Hageman GJ, Van Deun K, van den Hurk C, van Eenbergen M, Mols F; PROFILES Registry Group. Measuring Clinical, Biological, and Behavioral Variables to Elucidate Trajectories of Patient-Reported Outcomes: The PROFILES Registry. J Natl Cancer Inst. 2022 Jun 13;114(6):800-807. doi: 10.1093/jnci/djac047. PMID 35201353
- [Derived] van de Graaf DL, Mols F, Trompetter HR, van der Lee ML, Schreurs KMG, Borosund E, Nes LS, Smeets T. Effectiveness of the online Acceptance and Commitment Therapy intervention "Embrace Pain" for cancer survivors with chronic painful chemotherapy-induced peripheral neuropathy: study protocol for a randomized controlled trial. Trials. 2022 Aug 9;23(1):642. doi: 10.1186/s13063-022-06592-3. PMID 35945582
- See also: Data security and data access — http://www.profilesregistry.nl